CLINICAL TRIAL: NCT05215314
Title: Neurobiological Mechanisms of Perceived Stress and Their Modification Through Behavioral Intervention
Brief Title: Brain and Meditation (BAM) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1109; Protocol Version 10/12/2022 (Other: UW Madison); A483000 (Other: UW Madison); 5K01MH117222 (NIH)
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Stress; Behavior
Keywords: healthy minds program; mobile health
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Minds Program (HMP) (Experimental): Fully remote, 4-week meditation intervention
  Interventions: Behavioral: mHealth Meditation
- Waitlist Control (No Intervention): Control participants will not complete the Healthy Minds Program during the study, but can use it after they have completed the study

INTERVENTIONS:
Behavioral: mHealth Meditation — Participants will receive access to the 4-week Healthy Minds Program (HMP) Foundations module. The HMP app is a meditation-based smartphone app designed to promote and protect psychological well-being through sustainable skills training. The program is grounded in constituents of psychological well-being identified in empirical literature. HMP provides core content, with instruction administered through a curriculum of guided practices. HMP is based on research on eudaimonic well-being (e.g., environmental mastery, purpose) and brain-based skills that underlie these qualities (e.g., regulation of attention, mental flexibility). The full HMP has guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose. At post-treatment, participants will be given access to additional HMP content to support their continued practice.
  Other Names: mobile health app
  Arms: Healthy Minds Program (HMP)

SUMMARY:
This study is a randomized controlled trial to test the impact of an app-based meditation program on perceived stress and behavioral correlates of stress with known neurobiological correlates. Healthy adult participants between the ages of 25-65 will be enrolled in the study for about 4-5 months.

DETAILED DESCRIPTION:
Participants will be randomized into one of two groups: the intervention group or the waitlist control group. The intervention group will use a mobile health app for four weeks. Participants will complete pre-intervention, weekly, post-intervention, and 3-month follow-up surveys and tasks.

Primary Objective: Test for hypothesized group differences in perceived stress during participation in a 4-week meditation program and at 3-month follow-up.

Secondary Objective: Within the meditation group, determine whether reductions in perceived stress are associated with changes in hippocampal-dependent behavior.

ELIGIBILITY:
Inclusion Criteria:

* Individual can read, write, speak, and understand English
* Able to provide informed consent
* Willing and able to complete all study procedures, including the Healthy Minds Program
* Has access to a smartphone that can download apps from Google Play or the Apple App Store
* US citizen or a permanent US resident (green card holder)

Exclusion Criteria:

* Extensive experience in meditation practice (e.g., regular daily meditation practice for the past 6 months or regular weekly meditation practice for the past 12 months), experience in substantively similar meditation training programs (e.g., attended a meditation retreat or a yoga/body practice retreat with a significant mediation component), or substantial previous use of the Healthy Minds Program app
* Individuals will be excluded if they previously participated in substantively similar research at our Center at the discretion of the investigator due to similar tasks being used in certain studies
* History of psychosis
* History of mania
* Current psychopathology that interferes with study participation

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Grupe, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Center for Healthy Minds, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators may share coded data with researchers to address future research questions not included in this application, with a complementary study being conducted at the Center for Healthy Minds which is utilizing many of the same survey and behavioral task measures, and/or with journals where open data sharing policies are encouraged or are a requirement for publication. Coded data may be shared as Supplemental Information uploaded to journal websites.
  The investigators may share fully de-identified data from the study on data sharing platforms (e.g., OSF, NIMH Data Archive) for use by non-collaborators. Data shared on data sharing platforms will be uploaded via the internet. Confidentiality will be protected by stripping the data of all identifiers, including HIPAA identifiers.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Heller AS, Shi TC, Ezie CEC, Reneau TR, Baez LM, Gibbons CJ, Hartley CA. Association between real-world experiential diversity and positive affect relates to hippocampal-striatal functional connectivity. Nat Neurosci. 2020 Jul;23(7):800-804. doi: 10.1038/s41593-020-0636-4. Epub 2020 May 18. PMID 32424287

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Minds Program (HMP) | Waitlist Control
Started | 100 | 50
Completed | 95 | 48
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Minds Program (HMP) | Waitlist Control | Total
Number analyzed (Participants) | 100 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (10) | 40.6 (11) | 40.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 25 | 75
  Male | 50 | 25 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 21
  Not Hispanic or Latino | 86 | 42 | 128
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 10 | 22
  White | 70 | 27 | 97
  More than one race | 8 | 6 | 14
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 100 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Change in Perceived Stress Scale (PSS) Score
Description: PSS is a 10-item survey scored on a 5 point likert scale from 0 = never to 4 = very often, for a total possible range of scores from 0-40 where higher scores indicate higher perceived stress.
Time Frame: Baseline, following week 1, week 2, week 3, week 4 of intervention period, and 3 month follow-up
Population: The number analyzed changes over time because not all participants provided complete data for this measure at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) | Waitlist Control
Number analyzed (Participants) | 99 | 50
score on a scale
  baseline | 15.0 (6.49) | 17.1 (7.42)
  week 1: number analyzed (Participants) | 96 | 50
  week 1 | 13.5 (6.71) | 17.1 (7.48)
  week 2: number analyzed (Participants) | 94 | 48
  week 2 | 13.1 (7.03) | 15.1 (7.94)
  week 3: number analyzed (Participants) | 94 | 49
  week 3 | 12.5 (6.43) | 15.6 (6.52)
  week 4: number analyzed (Participants) | 94 | 49
  week 4 | 13.6 (6.6) | 16.7 (6.91)
  3 month follow up: number analyzed (Participants) | 95 | 48
  3 month follow up | 13.8 (6.96) | 17.8 (6.76)

2. Secondary Outcome: Change in Behavioral Pattern Separation Task
Description: Participants will complete a behavioral pattern separation task . During this task, participants will encode pictures of common objects while performing a basic categorization task. Participants will then label pictures as "Old" (targets, identical objects to those in the encoding phase), "New" (foils, or completely novel objects), or "Similar" (lure items, distinct exemplars of objects seen during encoding). The measure of interest on this task is the "Lure Discrimination Index", which is calculated as the proportion of lures correctly identified as "similar" minus the proportion of foils that are incorrectly identified as "similar". The theoretical range for the pattern separation index is [-1,1], with higher scores indicating better performance.
Time Frame: Baseline, following week 4 of intervention period, and 3 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Lure Discrimination Index
Arm/Group | Healthy Minds Program (HMP) | Waitlist Control
Number analyzed (Participants) | 94 | 47
Lure Discrimination Index
  baseline: number analyzed (Participants) | 94 | 46
  baseline | .507 (.201) | .456 (.197)
  week 4: number analyzed (Participants) | 85 | 45
  week 4 | .502 (.212) | .489 (.179)
  3 month follow up: number analyzed (Participants) | 91 | 47
  3 month follow up | .542 (.169) | .483 (.205)

3. Secondary Outcome: Change in PROMIS Depression Score
Description: The PROMIS Depression Score is a measure of feelings of depression in the past 7 days. This is a computer-adaptive survey scored on a 5 point likert scale from 1 (never) to 5 (always) with higher scores indicating increased depression. For analysis, total scores will be converted to t scores with a mean of 50 and SD of 10. Higher t scores indicate higher levels of depression. A t score >= 59.9 is indicative of moderate depression, a t score >= 65.8 is indicative of moderately severe depression, and a t score >= 71.5 is indicative of severe depression (based on corresponding cutoffs on the Patient Health Questionnaire-9).
Time Frame: Baseline, following week 1, week 2, week 3, week 4 of intervention period, and 3 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) | Waitlist Control
Number analyzed (Participants) | 99 | 50
score on a scale
  baseline | 52.4 (7.16) | 54.7 (7.28)
  week 1: number analyzed (Participants) | 96 | 50
  week 1 | 51.6 (8.17) | 54.8 (7.42)
  week 2: number analyzed (Participants) | 94 | 48
  week 2 | 51.3 (8.08) | 42.3 (9.28)
  week 3: number analyzed (Participants) | 94 | 49
  week 3 | 51.1 (8.27) | 55.0 (8.35)
  week 4: number analyzed (Participants) | 94 | 49
  week 4 | 50.2 (7.97) | 52.8 (8.25)
  3 month follow up: number analyzed (Participants) | 95 | 48
  3 month follow up | 51.9 (8.44) | 54.4 (7.91)

4. Secondary Outcome: Change in PROMIS Anxiety Score
Description: The PROMIS Anxiety Score is a measure of feelings of anxiety in the past 7 days. This is a computer-adaptive survey scored on a 5 point likert scale from 1 (never) to 5 (always) with higher scores indicating increased anxiety. For analysis, total scores will be converted to t scores with a mean of 50 and SD of 10. Higher t scores indicate higher levels of anxiety. A t score >= 62.3 is indicative of moderate anxiety and a t score >= 67.7 is indicative of severe anxiety (based on corresponding cutoffs on the General Anxiety Disorder-7).
Time Frame: Baseline, following week 1, week 2, week 3, week 4 of intervention period, and 3 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) | Waitlist Control
Number analyzed (Participants) | 99 | 50
score on a scale
  baseline | 55.8 (7.36) | 58.0 (8.46)
  week 1: number analyzed (Participants) | 96 | 50
  week 1 | 55.3 (7.56) | 57.4 (8.31)
  week 2: number analyzed (Participants) | 94 | 48
  week 2 | 54.9 (8.05) | 55.8 (7.70)
  week 3: number analyzed (Participants) | 94 | 49
  week 3 | 54.0 (7.95) | 57.4 (7.90)
  week 4: number analyzed (Participants) | 94 | 49
  week 4 | 53.1 (8.30) | 56.2 (8.72)
  3 month follow up: number analyzed (Participants) | 95 | 48
  3 month follow up | 54.3 (8.06) | 57.5 (6.94)

5. Other Pre Specified Outcome: Change in Posttraumatic Stress Disorder Checklist (PCL-5) Score
Description: The PCL-5 is a 20-item survey scored on a 5 point likert scale from 0 (not at all) to 4 (extremely) for a total possible range of score from 0-80 where higher scores indicate more symptoms of PTSD within the last 30 days.
Time Frame: Baseline, following week 4 of intervention period, and 3 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) | Waitlist Control
Number analyzed (Participants) | 99 | 50
score on a scale
  Baseline | 15.6 (12.2) | 17.2 (13.0)
  week 4: number analyzed (Participants) | 94 | 49
  week 4 | 13.2 (12.1) | 17.8 (16.1)
  3-month follow-up: number analyzed (Participants) | 95 | 48
  3-month follow-up | 13.9 (12.6) | 20.1 (13.4)

6. Other Pre Specified Outcome: Change in PROMIS Sleep Disturbance Score
Description: The PROMIS Sleep Disturbance Score is a measure of sleep in the past 7 days. This is a computer-adaptive survey scored on a 5 point likert scale with higher scores indicating increased sleep disturbance. For analysis, total scores will be converted to t scores with a mean of 50 and SD of 10. Higher t scores indicate higher levels of sleep disturbances. A t score >= 45.1 is indicative of significant sleep disturbances (based on a corresponding cutoff of >= 5 on the Pittsburgh Sleep Quality Index).
Time Frame: Baseline, following week 1, week 2, week 3, week 4 of intervention period, and 3 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) | Waitlist Control
Number analyzed (Participants) | 99 | 50
score on a scale
  Baseline | 52.0 (8.12) | 54.4 (9.28)
  week 1: number analyzed (Participants) | 96 | 50
  week 1 | 51.3 (9.05) | 54.0 (9.24)
  week 2: number analyzed (Participants) | 94 | 48
  week 2 | 50.6 (8.27) | 52.9 (9.66)
  week 3: number analyzed (Participants) | 94 | 49
  week 3 | 49.8 (9.33) | 53.6 (8.92)
  week 4: number analyzed (Participants) | 94 | 49
  week 4 | 50.1 (9.10) | 53.3 (9.95)
  3-month follow-up: number analyzed (Participants) | 95 | 48
  3-month follow-up | 50.5 (8.60) | 55.1 (9.84)

7. Other Pre Specified Outcome: Change in Five-facet Mindfulness Questionnaire: Awareness Subscale (FFMQ-A8) Score
Description: The FFMQ-A8 is an 8-item survey scored on a 5 point likert scale from 'never, or very rarely true' to 'very often or always true', for a total possible range of scores from 8-40 where higher scores indicate greater mindfulness awareness.
Time Frame: Baseline, following week 4 of intervention period, and 3 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) | Waitlist Control
Number analyzed (Participants) | 99 | 50
score on a scale
  Baseline: number analyzed (Participants) | 99 | 49
  Baseline | 27.9 (6.88) | 27.8 (7.36)
  week 4: number analyzed (Participants) | 94 | 50
  week 4 | 28.3 (6.02) | 28.3 (7.41)
  3-month follow-up: number analyzed (Participants) | 95 | 48
  3-month follow-up | 29.1 (6.41) | 28.0 (7.41)

8. Other Pre Specified Outcome: Change in NIH Toolbox Loneliness Score
Description: NIH toolbox Loneliness is a 5-item survey scored on a 5 point likert scale. The average score is taken across items for a total possible range of scores from 1-5, where higher scores indicate increased loneliness.
Time Frame: Baseline, following week 4 of intervention period, and 3 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) | Waitlist Control
Number analyzed (Participants) | 99 | 50
score on a scale
  Baseline | 2.44 (1.02) | 2.28 (0.84)
  week 4: number analyzed (Participants) | 94 | 49
  week 4 | 2.17 (1.00) | 2.19 (0.90)
  3-month follow-up: number analyzed (Participants) | 95 | 48
  3-month follow-up | 2.25 (1.07) | 2.25 (0.95)

9. Other Pre Specified Outcome: Change in Healthy Minds Index (HMI) Score
Description: HMI is a 17-item survey scored on a 5 point likert scale from 0 (never, none, not at all) to 4 (always, every time, to the highest degree) that assesses awareness, connection, insight, and purpose. Higher scores indicate higher sense of awareness, connection, insight, and purpose. Mean score for each subscale will be reported.
Time Frame: Baseline and following week 4 of intervention period
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Roaming Entropy
Description: Roaming entropy will be calculated according to the formula in Heller et al. (2020). Using continuous GPS location tracking, the measure takes into account distance traveled and distinct locations visited, with a single resulting value reflecting the diversity of movement through one's lived environment (Measured continuously throughout study participation)
Time Frame: Exploratory analyses will examine linear and nonlinear trajectories of change from baseline through 3-month follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 5 months (between enrollment and follow-up data completion)
Description: Definitions do not differ from those on clinicaltrials.gov
Arm/Group | Healthy Minds Program (HMP) | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/50
Other Adverse Events (participants affected / at risk) | 0/99 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT05215314/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT05215314/ICF_001.pdf